CLINICAL TRIAL: NCT05412862
Title: A Novel Psychological-behavioral Intervention to Promote Physical Activity After Acute Coronary Syndrome
Brief Title: Positive Emotions Following Acute Cardiac Events
Acronym: PEACE-V
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Director, Cardiac Psychiatry Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P003302
Record Dates: First submitted 2022-05-25; First posted 2022-06-09 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Acute Coronary Syndrome; Physical Inactivity
Keywords: Positive psychology; Physical Activity; Motivational Interviewing; Adherence
MeSH Terms: conditions — Acute Coronary Syndrome; Sedentary Behavior; Motor Activity | interventions — Psychology, Positive; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Randomized, single-blinded, controlled trial
Who Masked: Outcomes Assessor
Masking Description: Participants and treating study staff will be aware of the participant's treatment condition. However, follow-up assessments will be performed by a study staff member that is masked to the participant's treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology + Motivational Interviewing (Experimental): Each week, participants in the PP-MI intervention group will complete a PP activity and work towards a physical activity goal, then complete a phone session with a study trainer. Each phone session will include PP and goal setting portions. In the PP portion, the study trainer will (a) review the week's PP exercise, (b) discuss the rationale of the next week's PP exercise through a guided review of the PP-MI manual, and (c) assign the next week's PP exercise. In the goal-setting portion, the trainer will (a) review the participant's physical activity goal from the prior week, (b) discuss techniques for improving physical activity (e.g. tracking activity), and (c) help the participant to set a physical activity goal for the next week. Participants also will receive supplemental text messages throughout the 12 weeks of the intervention and during the initial follow-up period (Week 13-24).
  Interventions: Behavioral: Positive Psychology + Motivational Interviewing
- Treatment as Usual (No Intervention): Participants in the treatment as usual (TAU) arm will not receive any specific intervention, though they will be free to receive any post-ACS treatment.

INTERVENTIONS:
Behavioral: Positive Psychology + Motivational Interviewing — The 12-week PP-MI intervention focuses on enhancing well-being (through PP) and increasing physical activity (through MI). Each week, participants will complete a PP activity and work towards a physical activity goal, then complete a phone session with a study trainer. The PP portion of the program will focus on the cultivation of well-being through the performance of easy-to complete activities (e.g., using a strength in a new way) and review of the positive feelings they generate. The MI portion of the program will focus on assisting participants to improve physical activity levels, resolve ambivalence to behavior change, set realistic physical activity goals, problem-solve barriers, and identify resources to complete behavior change. Finally, participants will receive twice weekly text messages (for 24 weeks) to encourage completion of PP activities and engagement in physical activity.
  Arms: Positive Psychology + Motivational Interviewing

SUMMARY:
The focus of this study is to test the efficacy of a 12-week, remotely delivered, positive-psychology-motivational interviewing (PP-MI) intervention, with additional twice weekly text messages for a total of 24 weeks (with interactive, algorithm-driven, goal-focused text messages in the final 12 weeks), compared to post-acute coronary syndrome (ACS) treatment as usual, in a randomized trial of 280 post-ACS patients with low baseline physical activity.

DETAILED DESCRIPTION:
The investigators are proposing a study that will focus on testing the efficacy of a PP-MI intervention, with additional twice text messages for a total of 24 weeks (with interactive, algorithm-driven, goal-focused text messages in the final 12 weeks) in post-ACS patients. The investigators will enroll 280 post-ACS patients, who will take part in either a 12-week intervention (with 24 weeks of supplemental text messages), or receive post-ACS treatment as usual.

In this project, the investigators hope to do the following:

1. Examine the efficacy of a 12-week, phone-delivered PP-MI intervention for individuals with ACS on physical activity-related outcomes, as compared to the treatment as usual group.
2. Assess the intervention's impact on psychological (e.g. positive affect), functional (e.g. physical function), and behavioral (e.g. overall adherence) outcomes.
3. Explore the intervention's impact on markers of cardiovascular health (e.g., cardiac biomarkers), as well as major adverse cardiac events/readmissions.

Participants will be screened and enrolled during admission for an ACS. They will be provided with a accelerometer to monitor their physical activity for one week prior to their first in-person visit. At their first visit, they will answer questionnaires related to psychological and physical health and functioning, have their blood pressure and weight measured, and provide a fasting blood sample. Upon confirmation of adequate physical activity, participants will be randomized to receive the PP-MI intervention or treatment as usual.

Participants in the intervention will be provided a treatment manual, an activity tracker, and other treatment materials. The intervention will be introduced, and the first exercise will be assigned.

Following the first in-person visit, participants in the treatment condition will complete twelve weekly phone sessions with a study trainer. The phone sessions primarily will include a review of the prior week's session content and a discussion of the rationale and assignment of the next week's exercise/assignment.

Participants in the treatment condition will receive twice weekly text messages throughout the intervention (Weeks 1-12) and initial follow-up period (Weeks 13-24). These messages will focus on the PP activity and physical activity. During Weeks 13-24, participants in the PP-MI condition will engage with twice weekly, automated, interactive text messages related to PP and physical activity.

At Weeks 12, 24, and 48, participants will complete follow-up visits. One week prior to these visits, participants will be mailed an accelerometer and will wear it until their study visit. During these study visits, participants will be asked to answer questionnaires related to psychological and physical health and functioning, have their blood pressure and weight measured, and be asked about cardiovascular outcomes, including hospitalizations, cardiovascular procedures, and cardiac-specific hospitalizations. They will also provide a fasting blood sample.

Finally, participants will complete phone sessions every 6 months until study end to inquire about hospitalizations and adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* ACS (myocardial infarction or unstable angina)
* Suboptimal physical activity (score of < 6 on the Medical Outcomes study Specific Adherence Scale item related to physical activity)

Exclusion Criteria:

* Cognitive deficits (assessed via a 6-item cognitive screening tool)
* Medical conditions likely to lead to death within 6 months.
* Moderate-severe depression (Patient Health Questionnaire-9 [PHQ-9] score ≥15)
* Inability to participate in physical activity due to another medical condition (e.g., arthritis)
* Inability to read, write, or speak in English
* Inability to receive text-messages
* Current participation in another intervention or program that has been designed to promote well-being or physical activity

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Moderate to Vigorous Physical Activity (MVPA) at 24 weeks | Measured for 7 days at baseline and 24 weeks
  MVPA will be measured via an accelerometer and recorded in mean minutes/day.

SECONDARY OUTCOMES:
Change in Light Intensity Activity | Measured for 7 days at baseline, 12 weeks, 24 weeks, and 48 weeks
  Light intensity activity will be measured via an accelerometer and recorded in mean minutes/day.
Change in positive affect (Positive and Negative Affect Schedule [PANAS] positive affect items) | Baseline, 12 weeks, 24 weeks, 48 weeks
  The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials and in patients with HF, will be used to measure positive affect (Range: 10-50). Higher scores indicate higher levels of positive affect.

OTHER OUTCOMES:
Change from Baseline Moderate to Vigorous Physical Activity (MVPA) at 12 and 48 weeks | Measured for 7 days at baseline, 12 weeks, and 48 weeks
  MVPA will be measured via an accelerometer and recorded in mean minutes/day.
Change in Sedentary time | Measured for 7 days at baseline, 12 weeks, 24 weeks, and 48 weeks
  Sedentary time will be measured via an accelerometer and recorded in mean minutes/day.
Change in optimism (Life Orientation Test - Revised [LOT-R]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Life Orientation Test-Revised (LOT-R) is a well-validated 6-item instrument used to measure dispositional optimism (Range: 0-24). Higher scores indicate higher levels of dispositional optimism.
Change in depressive symptoms (Patient Health Questionnaire [PHQ-9]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  The Patient Health Questionnaire-9 (PHQ-9) will be used to measure depression. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-27). Higher scores indicate higher levels of depression.
Change in anxiety (Hospital Anxiety and Depression Scale - anxiety subscale [HADS-A]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  The Hospital Anxiety and Depression Scale (HADS)-anxiety subscale will be used to measure anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients (Range: 0-21). Higher scores indicate higher levels of anxiety.
Change in locus of control (Form C of the Multidimensional Health Locus of Control scale [MHLC Form C]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Locus of control will be measured using the 18-item Multidimensional Health Locus of Control scale [MHLC Form C]. Scores on this scale range from 6-36, with higher scores indicating greater internal health locus of control.
Change in perceived social support (Multidimensional Scale of Perceived Social Support [MSPSS]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  The MSPSS is a 12-item scale designed to measure perceived social support from three sources: Family, Friends, and a Significant Other. Scores on this scale range from 0-84, with higher scores indicating greater perceived social support.
Change in exercise-related self-efficacy (Self-efficacy for Exercise Scale [SEE]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  The Self-efficacy for Exercise Scale will be used to measure exercise self-efficacy. This is a 9-item scale used to assess an individual's beliefs in their ability to continue exercising on a three time per week basis at moderate intensities for 20+ minutes per session in the future. Scores on this scale range from 0-90, with higher scores indicating greater self-efficacy for exercise.
Change in physical function (PROMIS 20-item Physical Function Short Form [PF-20]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  The PROMIS 20-item short form (PF-20) will be used to assess physical function. Scores on this scale range from 20-100, with higher scores indicating greater physical function.
Change in mental health-related quality of life(Medical Outcomes Study Short Form-12 [SF-12] mental component score) | Baseline, 12 weeks, 24 weeks, 48 weeks
  The SF-12 mental component score will be used to assess mental health-related quality of life (Range: 0-100). Higher scores indicate higher levels of mental health-related quality of life.
Change in physical health-related quality of life (Medical Outcomes Study Short Form-12 [SF-12] physical component score) | Baseline, 12 weeks, 24 weeks, 48 weeks
  The SF-12 physical component score will be used to assess physical health-related quality of life (Range: 0-100). Higher scores indicate higher levels of physical health-related quality of life.
Change in adherence to cardiac medications | Baseline, 12 weeks, 24 weeks, 48 weeks
  Medication adherence will be measured with the self-report medication adherence tool from the NHLBI Heart and Soul Study.
Change in Fat/saturated fat/cholesterol intake (Meat, Eggs, Dairy, Fried foods, fat In baked goods, Convenience foods, fats added at the Table, and Snacks [MEDFICTS]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Measured by the MEDFICTS scale, a National Cholesterol Education Program-developed scale inquiring about saturated fat.
Change in self-reported MVPA (International Physical Activity Questionnaire [IPAQ]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Measured by the self-report International Physical Activity Questionnaire (IPAQ). The measure assesses the types of intensity of physical activity that people do as part of their daily lives. Moderate and vigorous intensity activities will be converted to multiples of resting energy expenditure (MET) minutes per week.
Change in self-reported sedentary time (International Physical Activity Questionnaire [IPAQ]) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Measured by the self-report International Physical Activity Questionnaire (IPAQ). Measured in hours per day.
Major adverse cardiac events (MACE) | Through study completion, an average of 2.7 years
  MACE will be defined as mortality or hospitalization for heart failure or an acute coronary event (percutaneous coronary intervention or acute coronary syndrome). Data regarding hospitalizations and mortality will be obtained using a three-pronged approach consisting of systematic queries of participants, electronic health record review, and review of records from the National Death Index.
All-cause hospitalizations | Through study completion, an average of 2.7 years
  We will record all-cause hospitalizations for all participants from enrollment to the end of the study data collection period, using systematic queries of participants and review of electronic health records from all Mass General Brigham-affiliated hospitals.
Attendance at cardiac rehabilitation | 12 weeks, 24 weeks, 48 weeks
  We will query participants at each follow-up time point to determine whether they have attended cardiac rehabilitation.
Change in weight (kilograms) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Weight will be measured during study visits.
Change in body mass index (kilograms per square meter) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Height and weight will be measured during study visits.
Change in blood pressure (millimeters of mercury) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Blood pressure (diastolic and systolic) will be measured by trained nurses using a standardized protocol.
Change in low density lipoprotein (LDL) and high density lipoprotein (HDL) cholesterol (milligrams per deciliter) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Fasting blood samples will be obtained at study visits.
Change in triglycerides (milligrams per deciliter) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Fasting blood samples will be obtained at study visits.
Change in glucose (milligrams per deciliter) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Fasting blood samples will be obtained at study visits.
Change in interleukin-6 (picograms per milliliter) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Blood samples will be obtained at study visits.
Change in high sensitivity C-reactive protein (milligrams per liter) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Blood samples will be obtained at study visits.
Change in endothelin-1 (picograms per milliliter) | Baseline, 12 weeks, 24 weeks, 48 weeks
  Blood samples will be obtained at study visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff C Huffman, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
To promote sharing of study data with other researchers, we will create a deidentified study dataset. We will include both item-level and summary scores for each scale and will include data from the baseline, 12-week, 24-week, and 48-week time points.
Supporting Information: Study Protocol, SAP
Time Frame: This information will be shared prior to the end of the study funding period.
Access Criteria: Investigators who are interested in obtaining access to this information will be asked to submit a request to the principal investigator outlining the proposed use of the data and would need to agree to certain conditions (e.g., not attempting to identify individual participants, destroying data once the use of the data is complete) prior to obtaining access.